CLINICAL TRIAL: NCT03506893
Title: Medical-economic Evaluation of the Care of Refractory Ascites by Implantation of Alfapump® Device in Cirrhotic Patients
Acronym: ARIAPUMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.109
Record Dates: First submitted 2018-03-08; First posted 2018-04-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Ascites; Paracentesis; Cirrhosis
Keywords: refractory ascite; pump system
MeSH Terms: conditions — Ascites; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alphapump (Experimental): Alfapump® device implantation under general anesthesia (30-45 minutes)
  Interventions: Device: Alphapump
- Ascites puncture (Active Comparator): Iterative paracentesis compensated for by albumin infusions in ambulatory care.
  Interventions: Procedure: Ascites puncture

INTERVENTIONS:
Device: Alphapump — Alfapump® device: a completely internalized medical device, implanted under the skin, which mobilizes ascites from the peritoneal cavity to the bladder where they are eliminated by the urinary tract.
  Medical device marked CE, used in the indication provided for marking
  Arms: Alphapump
Procedure: Ascites puncture — Hospitalizations for evacuating ascites are performed at least twice a month and can be up to 2 times a week. A clinical and biological examination is carried out at each visit.
  Arms: Ascites puncture

SUMMARY:
The hypothesis is that the Alfapump® strategy would be more effective in terms of QALYs generated , and that the cost of Alfapump® device and its implantation will be totally or partially offset by the reduction in the number of evacuating parentheses performed and the reduction in the number of complications in patients with refractory ascites awaiting liver transplantation or not. On the other hand, given the difference in the clinical profiles of these two populations (whether or not they are awaiting transplantation), these two populations will be study separately

Evaluation of the medical-economic impact at 1 year of the two therapeutic strategies: implantation of Alfapump® versus repeated evacuating paracentesis in cirrhotic patients with refractory ascites without scheduled liver transplantation.

DETAILED DESCRIPTION:
Refractory ascites is one of the complications associated with portal hypertension in the cirrhotic patient. To date, its treatment consists of evacuating punctures, performed in day hospitalisation, whose frequency is adapted to the rate of ascites synthetis. Paracentesis, which does not affect the mechanisms of ascites formation, contributes to protein catabolism and undernutrition. They also have an inconvenience linked to the gesture, making frequent hospital stays necessary. For all these reasons, the patient's quality of life is diminished. The Alfapump® system is a new method for the treatment of refractory ascites. It is a completely internalized medical device, implanted under the skin, which mobilizes ascites from the peritoneal cavity to the bladder, where ascites is eliminated by urinary tract.

ELIGIBILITY:
Inclusion Criteria:

* Patient with refractory ascites who has had a minimum of 5 paracentesis in the last 3 months.
* Patient with an estimated life expectancy of at least 6 months on the day of inclusion.
* Patient with contraindication to the application of a TIPS or who has expressed a refusal of the procedure or a non-functional TIPS
* Patient affiliated with or in receipt of social security
* Informed and written consent signed by the patient.

Exclusion Criteria:

* Local or systemic infection in the month preceding the procedure
* Hepatocellular carcinoma with palliative care
* MELD Score > 18
* Child Pugh C Score > 10
* Creatinine Clearance < 50 ml/mn
* Digestive hemorrhage or episode of hepatic encephalopathy within two weeks prior to device insertion
* Contraindication to general anesthesia
* Contraindication to implant surgery of the device:

  * Obstructive urological impairment
  * Partitioning of ascites
  * Coagulopathy
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant woman, parturient, breastfeeding mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure).
* Patient currently participating in other clinical research or who participated in a clinical trial within one month prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of medical-economic impact at 1 year of 2 strategies: implantation of Alfapump® device versus repeated evacuating paracentesis (reference treatment) in cirrhotic patients with refractory ascites without programmed liver transplantation. | 1 year
  Incremental cost-utility ratio (ICER) from societal perspective.

SECONDARY OUTCOMES:
Comparison of the clinical impact at 6 and 12 months of Alfapump® versus repeated evacuating paracentesis in cirrhotic patients with refractory ascites WITHOUT programmed liver transplantation. | 6 months and 1 year
  Evaluation of the paracentesis-free survival, cirrhosis and device-related adverse events.
Evaluation of the clinical impact at 6 and 12 months of Alfapump® versus repeated evacuating paracentesis in cirrhotic patients with refractory ascites WITH programmed liver transplantation. | 6 months and 1 year
  Evaluation of the paracentesis-free survival, cirrhosis and device-related adverse events.
Evaluation of the economic impact at 6 and 12 months of Alfapump® versus repeated evacuating paracentesis in cirrhotic patients with refractory ascites WITH programmed liver transplantation. | 6 months and 1 year
  Incremental cost-utility ratio.
Evaluation of the clinical impact at 2 years of Alfapump® versus repeated evacuating paracentesis (prospective observational study). | 2 years
  Evaluation of paracentesis-free survival, cirrhosis and device-related adverse events. We will analyse separately patients WITH and WITHOUT programmed liver transplantation.
Evaluation of the economic impact at 2 years of Alfapump® versus repeated evacuating paracentesis (prospective observational study). | 2 years
  Incremental cost-utility ratio. We will analyse separately patients WITH and WITHOUT programmed liver transplantation.
Budget impact Analysis from the point of view of French health insurance, at 3 and 5 years. | 3 and 5 years
  Economic consequences of the introduction of the Alfapump® device in the management strategies of cirrhotic patients presenting a refractory ascites.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Noelle HILLERET, MD, Principal Investigator — University Hospital, Grenoble
Locations (10):
- France (10):
  - Amiens-Picardie University Hospital, Amiens
  - Chu Angers, Angers
  - Jean MINJOZ Univesity Hospital, Besançon
  - Haut-Lévêque Hospital, Bordeaux
  - Beaujon Hospital, Clichy
  - Grenoble University Hospital, Grenoble
  - LA PITIE SALPETRIERE Univesity Hospital, Paris
  - Chu Poitiers, Poitiers
  - Chu Pontchaillou, Rennes
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellot P, Welker MW, Soriano G, von Schaewen M, Appenrodt B, Wiest R, Whittaker S, Tzonev R, Handshiev S, Verslype C, Moench C, Zeuzem S, Sauerbruch T, Guarner C, Schott E, Johnson N, Petrov A, Katzarov K, Nevens F, Zapater P, Such J. Automated low flow pump system for the treatment of refractory ascites: a multi-center safety and efficacy study. J Hepatol. 2013 May;58(5):922-7. doi: 10.1016/j.jhep.2012.12.020. Epub 2013 Jan 11. PMID 23318604
- [Background] Bureau C, Adebayo D, Chalret de Rieu M, Elkrief L, Valla D, Peck-Radosavljevic M, McCune A, Vargas V, Simon-Talero M, Cordoba J, Angeli P, Rosi S, MacDonald S, Malago M, Stepanova M, Younossi ZM, Trepte C, Watson R, Borisenko O, Sun S, Inhaber N, Jalan R. Alfapump(R) system vs. large volume paracentesis for refractory ascites: A multicenter randomized controlled study. J Hepatol. 2017 Nov;67(5):940-949. doi: 10.1016/j.jhep.2017.06.010. Epub 2017 Jun 21. PMID 28645737
- [Background] Stirnimann G, Berg T, Spahr L, Zeuzem S, McPherson S, Lammert F, Storni F, Banz V, Babatz J, Vargas V, Geier A, Stallmach A, Engelmann C, Trepte C, Capel J, De Gottardi A. Treatment of refractory ascites with an automated low-flow ascites pump in patients with cirrhosis. Aliment Pharmacol Ther. 2017 Nov;46(10):981-991. doi: 10.1111/apt.14331. Epub 2017 Sep 21. PMID 28940225
- [Background] Sola E, Sole C, Gines P. Management of uninfected and infected ascites in cirrhosis. Liver Int. 2016 Jan;36 Suppl 1:109-15. doi: 10.1111/liv.13015. PMID 26725907
- [Background] Thomas MN, Sauter GH, Gerbes AL, Stangl M, Schiergens TS, Angele M, Werner J, Guba M. Automated low flow pump system for the treatment of refractory ascites: a single-center experience. Langenbecks Arch Surg. 2015 Dec;400(8):979-83. doi: 10.1007/s00423-015-1356-1. Epub 2015 Nov 13. PMID 26566989
- [Background] Stepanova M, Nader F, Bureau C, Adebayo D, Elkrief L, Valla D, Peck-Radosavljevic M, McCune A, Vargas V, Simon-Talero M, Cordoba J, Angeli P, Rossi S, MacDonald S, Capel J, Jalan R, Younossi ZM. Patients with refractory ascites treated with alfapump(R) system have better health-related quality of life as compared to those treated with large volume paracentesis: the results of a multicenter randomized controlled study. Qual Life Res. 2018 Jun;27(6):1513-1520. doi: 10.1007/s11136-018-1813-8. Epub 2018 Feb 19. PMID 29460201